CLINICAL TRIAL: NCT05723263
Title: IGHID 12118 - Pay-it-forward Gonorrhea and Chlamydia Testing Among Men in China: The PIONEER Pragmatic Randomized Controlled Trial
Brief Title: Pay-it-forward Gonorrhea and Chlamydia Testing Among Men in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-1667; R01AI158826 (NIH)
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-03

CONDITIONS: Gonorrhea; Chlamydia
Keywords: gonorrhea; sexually transmitted infection (STI); gonorrhea testing among men who have sex with men; chlamydia
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: hybrid effectiveness-implementation study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Pay-it-forward (Experimental): * free gonorrhea/chlamydia testing
  * minimal engagement
  Interventions: Behavioral: Standard Pay-it-forward
- Community engaged Pay-it-forward (Experimental): * Free gonorrhea/chlamydia testing
  * Stronger engagement
  Interventions: Behavioral: Community Engaged Pay-it-forward
- Control arm (Other): * Test available for a fee
  * No engagement
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: Standard Pay-it-forward — 400 men who have sex with men (MSM) at 4 clinics will be enrolled. The standard pay-it-forward arm will include free point-of-care gonorrhea testing, as well as a passive community engagement component (such as viewing postcards and materials written by others encouraging gonorrhea/chlamydia testing).
  Arms: Standard Pay-it-forward
Behavioral: Community Engaged Pay-it-forward — 400 MSM at 4 clinics will be enrolled. The community engaged pay-it-forward arm will include free point-of-care gonorrhea testing, as well as an active community engagement component (such as multi-stakeholder co-creation activities to develop essential components of the intervention and implementation strategies; writing postcards; designing fans with stickers; sending out testing promotion messages on social media; and opportunity to donate to support others)
  Arms: Community engaged Pay-it-forward
Other: Control arm — 400 MSM at 4 clinics will be enrolled. The control arm will include a fee-based point-of-care gonorrhea testing (approximately 20 U.S. Dollars (USD) per test) and no community engagement component
  Arms: Control arm

SUMMARY:
PIONEER is a three-arm, programmatic cluster randomized controlled trial (RCT) to compare effectiveness of three implementation strategies, followed by a mixed-methods implementation evaluation study

DETAILED DESCRIPTION:
The study will be implemented at 12 clinics in Guangdong, China, which will be randomly assigned to one of the intervention arms for delivering gonorrhea testing: a standard pay-it-forward implementation strategy with minimal encouragement to get tested, a community-engaged pay-it-forward strategy, and a control arm in which men pay for their own sexually transmitted disease (STD) test. Data sources will include survey data on acceptability of intervention, intervention appropriateness, feelings and attitudes towards interventions among participants, administrative data about test uptake, treatment rate, and donations, as well as qualitative data to gain insights about men's perceptions and attitudes towards the pay-it-forward interventions strategies, mechanisms driving uptake and donating behaviors. Both survey and qualitative interviews with implementers and organizers about fidelity and adherence to protocol, intention to continue and maintain a pay-it-forward intervention, and barriers and facilitators of implementing the intervention will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* have had sex over the past year
* have not been tested for gonorrhea and chlamydia in the past year
* reside in the city in the past three months
* speak Mandarin Chinese or Cantonese
* mentally capable of providing informed consent to test for gonorrhea and chlamydia
* own a mobile phone

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tucker, MD, Principal Investigator — University of North Carolina
Locations (1):
- Dermatology Hospital, Institute for Global Health and Sexually Transmitted Diseases, Southern Medical University, China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Marley G, Tan RKJ, Wu D, Wang T, Sun M, Sheng Q, Holly ME, Hlatshwako TG, Wang C, Tang W, Ramaswamy R, Yang L, Luo D, Sylvia SS, Gray K, Van Duin D, Zheng H, Tucker JD. Pay-it-forward gonorrhea and chlamydia testing among men who have sex with men and male STD patients in China: the PIONEER pragmatic, cluster randomized controlled trial protocol. BMC Public Health. 2023 Jun 20;23(1):1182. doi: 10.1186/s12889-023-16095-8. PMID 37337181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referrals at six (6) public sexually transmitted infection (STI) and six (6) community-led clinics.
Pre-assignment Details: 12 clinics in six cities were randomized to the three intervention arms in a 1:1:1 ratio, stratified by the 2023 GDP ranking. Each city had two clinics, and all clinics in the same city were assigned to the same intervention arm.
  Of the 1312 participants screened, 1200 met inclusion criteria and received the intervention assigned to the clinic. Reasons for exclusion were as follows: tested for gonorrhea in the last 12 months = 111, and disagreed to provide informed consent = 1
Units Other Than Participants: Clinic randomization in 1:1:1 ratio
Groups:
- Community-Engaged Pay-It-Forward: Participants received free gonorrhea and chlamydia testing donated by previous participants and were offered an opportunity to make monetary and/or handwritten message donations to support other participants.
- Standard Pay-It-Forward: Participants received free gonorrhea and chlamydia testing donated by previous participants and were offered an opportunity to make monetary donations to support other participants.
- Control: Participants received gonorrhea and chlamydia testing at an out-of-pocket cost of approximately $21 U.S. Dollars (USD).
Period: Overall Study
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Started | 400; 4 Clinic randomization in 1:1:1 ratio | 400; 4 Clinic randomization in 1:1:1 ratio | 400; 4 Clinic randomization in 1:1:1 ratio
Completed | 400; 4 Clinic randomization in 1:1:1 ratio | 400; 4 Clinic randomization in 1:1:1 ratio | 400; 4 Clinic randomization in 1:1:1 ratio
Not Completed | 0; 0 Clinic randomization in 1:1:1 ratio | 0; 0 Clinic randomization in 1:1:1 ratio | 0; 0 Clinic randomization in 1:1:1 ratio

BASELINE CHARACTERISTICS:
Population: Men seeking HIV and STI care services at project public STI and community-led clinics.
Groups:
- Control: Participants received gonorrhea and chlamydia testing at an out-of-pocket cost of approximately $21 U.S.Dollars (USD).
- Total: Total of all reporting groups
Arm/Group | Community-engaged Pay-It-Forward | Standard Pay-It-Forward | Control | Total
Number analyzed (Participants) | 400 | 400 | 400 | 1200
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.36 (12.54) | 33.46 (12.49) | 34.90 (11.12) | 35.06 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 400 | 400 | 400 | 1200
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 400 | 400 | 400 | 1200
City of Enrollment [Count of Participants; unit: Participants]
  Dongguan | 0 | 0 | 200 | 200
  Foshan | 200 | 0 | 0 | 200
  Huizhou | 200 | 0 | 0 | 200
  Jiangmen | 0 | 200 | 0 | 200
  Zhanjiang | 0 | 0 | 200 | 200
  Zhuhai | 0 | 200 | 0 | 200
Marital Status [Count of Participants; unit: Participants]
  Ever Married | 201 | 133 | 190 | 524
  Never Married | 199 | 267 | 210 | 676
Sexual Behavior [Count of Participants; unit: Participants] — Self-reported history of anal sex with other men.
  Participants
    MSM | 194 | 230 | 197 | 621
    Non-MSM | 206 | 170 | 203 | 579
Highest Level of Education [Count of Participants; unit: Participants]
  Below high school | 118 | 87 | 80 | 285
  High school | 119 | 89 | 141 | 349
  Bachelor's degree | 136 | 186 | 130 | 452
  Postgraduate and above | 27 | 36 | 49 | 112
Annual Income [Count of Participants; unit: Participants] — United States Dollars (USD)
  Participants
    < $49,670 | 100 | 120 | 102 | 322
    $49,670 - $79,999 | 128 | 113 | 121 | 362
    >/= $80,000 | 172 | 167 | 177 | 516
Previous Testing [Count of Participants; unit: Participants] — Self-reported data on having ever tested for these sexually transmitted infections. Data was collected using a self-administered questionnaire at Baseline.
  Participants
    Gonorrhea | 58 | 51 | 35 | 144
    Chlamydia | 63 | 50 | 36 | 149

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Testing for Gonorrhea and Chlamydia
Description: Defined as the number of eligible participants who accepted and provided laboratory samples for gonorrhea and chlamydia PCR testing out of the total number of eligible participants recruited across the three study arms.
Time Frame: During enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 400
Participants | 390 | 361 | 12
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Control; It was calculated that 12 clinic sites with 1200 participants randomized in a 1:1:1 ratio between the three arms would have at least 90% power to detect a 10% difference in the proportion of test uptake between the pay-it-forward and control group participants, using a two-sided, two-sample t-test (α=0.05), assuming a 0.25~0.31 cluster coefficient of variation, a <5% lost-to-follow-up rate, and an intra-class correlation of 0.016; Test type: Other; p < 0.001, Generalized Estimating Equations — The threshold for statistical significance was p<0.05; Proportional difference = 94.5, 95% CI 2-sided [94.2 to 94.8]
Statistical Analysis 2: Comparison: Standard Pay-It-Forward vs Control; It was estimated that 12 clinic sites with 1200 participants randomized in a 1:1:1 ratio between the three arms would have at least 90% power to detect a 10% difference in the proportion of test uptake between the pay-it-forward and control group participants, using a two-sided, two-sample t-test (α=0.05), assuming a 0.25~0.31 cluster coefficient of variation, a <5% lost-to-follow-up rate, and an intra-class correlation of 0.016; Test type: Other; p < 0.001, Generalized Estimating Equations — The threshold for statistical significance was p<0.05; Proportional difference = 87.2, 95% CI 2-sided [86.5 to 88.0]
Statistical Analysis 3: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward; Using a binary outcome and cluster RCT design, we estimated that 12 clinic clusters (two per city) and 1200 participants (100 per cluster) were needed to achieve a 90% power and allow for a 0.05 type-I error to detect a 10% difference in the proportion of test uptake between the pay-it-forward and control arm participants and a <5% lost-to-follow-up rate. We anticipated a test uptake of 65% in the community-engaged pay-it-forward arm, 45% in the standard pay-it-forward arm, and 20% in control; Test type: Other; p > 0.05, Generalized Estimating Equations; Proportional difference = 7.3, 95% CI 2-sided [6.6 to 7.9]

2. Secondary Outcome: Donation Amount
Description: The response was defined as the total amount of money donated by participants in the pay-it-forward group to support testing for other participants. Self-reported via a self-administered survey and validated in donation receipt records.
Time Frame: Baseline
Population: Per-protocol population (all participants recruited to the community-engaged and standard pay-it-forward groups and offered a chance to donate). This outcome does not apply to participants in the Control arm.
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 0
USD | 225.16 (37.53) | 382.61 (63.77) |
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward; Test type: Other; p < 0.001, Chi-squared

3. Secondary Outcome: Number of Participants Who Test Positive for Gonorrhea
Description: The response rate was defined as the number of participants who tested positive for gonorrhea out of the total number of participants tested for gonorrhea. Test results were obtained from validated laboratory diagnosis reports based on polymerase chain reaction (PCR) testing.
Time Frame: Within 2 weeks of enrollment
Population: Per-protocol population (all participants tested for gonorrhea with laboratory results available).
Measure: Count of Participants; unit: Participants
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 390 | 361 | 12
Participants | 10 | 12 | 1
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; Test type: Other; p = 0.0059, Chi-squared

4. Secondary Outcome: Number of Participants Who Test Positive for Chlamydia
Description: The response rate was defined as the number of participants who tested positive for chlamydia out of the total number of participants who tested for chlamydia. Test results were obtained from validated laboratory diagnosis reports based on PCR testing.
Time Frame: Within 2 weeks of recruitment
Population: Per-protocol population (all participants tested for chlamydia with laboratory results available).
Measure: Count of Participants; unit: Participants
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 390 | 361 | 12
Participants | 35 | 58 | 0
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; Test type: Other; p < 0.001, Chi-squared

5. Secondary Outcome: Cost Per Test Per Individual
Description: The costs per test individual consist of the direct costs of PCR tests for gonorrhea and chlamydia for each individual tested at baseline. For the intervention arms, the estimate was calculated as the total direct cost paid to the laboratory minus the total amount donated by pay-it-forward arm participants in that intervention arm, divided by the total number of participants tested in that arm. The average exchange rate for the US dollar (USD) to RMB on March 31, 2025, was 1 USD = 7.22 RMB.
  Control arm participants paid the standard cost of 150 RMB (~20.18 USD) each for dual PCR testing at the clinic site out-of-pocket.
Time Frame: Baseline - During enrollment visit
Population: Per protocol analysis (cost of gonorrhea and chlamydia testing for each eligible participant who accepted and provided samples for dual gonorrhea and chlamydia testing in each study arm). Fraction for direct cost per test per individual = (total direct cost of laboratory tests paid - total amount donated by participants) / total number of participants tested.
Measure: Mean (Standard Deviation); unit: USD
Groups:
- Community Engaged Pay-it-forward: * Free gonorrhea/chlamydia testing
  * Stronger engagement
  Community Engaged Pay-it-forward: 400 MSM at 4 clinics will be enrolled. The community engaged pay-it-forward arm will include free point-of-care gonorrhea testing, as well as an active community engagement component (such as multi-stakeholder co-creation activities to develop essential components of the intervention and implementation strategies; writing postcards; designing fans with stickers; sending out testing promotion messages on social media; and opportunity to donate to support others)
- Standard Pay-it-forward: * free gonorrhea/chlamydia testing
  * minimal engagement
  Standard Pay-it-forward: 400 men who have sex with men (MSM) at 4 clinics will be enrolled. The standard pay-it-forward arm will include free point-of-care gonorrhea testing, as well as a passive community engagement component (such as viewing postcards and materials written by others encouraging gonorrhea/chlamydia testing).
- Control Arm: * Test available for a fee
  * No engagement
  Control arm: 400 MSM at 4 clinics will be enrolled. The control arm will include a fee-based point-of-care gonorrhea testing (approximately 20 U.S. Dollars (USD) per test) and no community engagement component
Arm/Group | Community Engaged Pay-it-forward | Standard Pay-it-forward | Control Arm
Number analyzed (Participants) | 390 | 361 | 12
USD | 14.10 (0.41) | 13.61 (0.75) | 20.18 (0)

6. Secondary Outcome: Mean Self Reported Gratitude Score
Description: The response rate was the average self-rated gratitude towards and about the pay-it-forward intervention. This was scored using a 10-item adapted gratitude survey on a 5-level Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Possible average scores ranged from 1 (lowest level of gratitude) to 7 (highest level of gratitude).
Time Frame: During enrollment visit
Population: Per-protocol population (all participants recruited to the pay-it-forward intervention group with average gratitude scores results available. Less than <15% missing data for items in this scale was observed and average imputation was used). This outcome does not apply to participants in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 0
score on a scale | 5.81 (1.04) | 6.21 (0.84) |
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward; Test type: Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Mean Self Reported Community Engagement Score
Description: The response rate was the average self-rated community engagement with the local and/or LGBTQ community before participating in the study, scored using a validated tool assessed on a 6-item Likert scale. Possible average scores ranged from 0 (no community engagement) to 6 (high community engagement)
Time Frame: Baseline
Population: Less than <15% missing data for items in this scale was observed and average imputation was used.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 400
score on a scale | 0.21 (0.29) | 0.27 (0.31) | 0.32 (0.34)
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; Test type: Other; p = 0.007, t-test, 2 sided

8. Secondary Outcome: Mean Community Connectedness and Cohesion Score
Description: The response rate was defined as the average self-rated community engagement score using a validated 11-item scale rated on a 4-level Likert scale. Possible average scores ranged from 1 (low community connectedness and cohesion) to 4 (high community connectedness and cohesion)
Time Frame: Baseline
Population: Per-protocol population (all participants with average community connectedness and cohesion score results available. Less than <15% missing data for items in this scale was observed and average imputation was used).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Arm: * Test available for a fee
  * No engagement
  Control arm: 400 MSM at 4 clinics will be enrolled. The control arm will include a fee-based point-of-care gonorrhea testing (approximately 20 USD per test) and no community engagement component
Arm/Group | Community Engaged Pay-it-forward | Standard Pay-it-forward | Control Arm
Number analyzed (Participants) | 400 | 400 | 400
score on a scale | 3.27 (0.67) | 3.02 (0.72) | 2.66 (0.83)
Statistical Analysis 1: Comparison: Community Engaged Pay-it-forward vs Standard Pay-it-forward vs Control Arm; Test type: Other; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Internalized Homophobia and Self-identification
Description: The response rate was the average self-rated internalized homophobia and self-identification score assessed using a validated 9-item survey rated on a 1-5 Likert scale. Possible average scores ranged from 1 (low self-identification and high internalized homophobia) to 5 (high self-identification and low internalized homophobia)
Time Frame: Baseline
Population: Per-protocol population (All MSM participants with internalized homophobia assessment results available. Less than <15% missing data for items in this scale was observed and average imputation was used). MSM referred to all eligible male participants who self-reported having ever engaged in anal intercourse with another man in the baseline survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community-Engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 194 | 230 | 197
score on a scale | 3.61 (0.89) | 3.34 (0.95) | 3.44 (0.84)
Statistical Analysis 1: Comparison: Community-Engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; Test type: Other; p = 0.727, t-test, 2 sided

10. Other Pre Specified Outcome: Gonorrhea and Chlamydia Testing Uptake by Clinic Type
Description: Stratifies gonorrhea/chlamydia testing uptake between participants recruited in community-led clinics versus public STI clinics across the three intervention arms.
Time Frame: During enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Community-engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 400
Participants
  Community-led Clinic | 199 | 164 | 1
  Public STI Clinic | 191 | 197 | 11
  Not Tested | 10 | 39 | 388
Statistical Analysis 1: Comparison: Community-engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; We anticipated a test uptake of 65% in the community-engaged pay-it-forward arm, 45% in the standard pay-it-forward arm, and 20% in the control between community-led and public STI clinic participants; Test type: Other; p = 0.005, Generalized Estimating Equations; Difference in Probability Difference = -0.047, 95% CI 2-sided [-0.080 to -0.014] — Absolute proportional difference in gonorrhea and chlamydia test uptake rate among community-led clinic participants across the three intervention arms

11. Other Pre Specified Outcome: Gonorrhea and Chlamydia Testing Uptake by Sexual Orientation
Description: Stratifies gonorrhea/chlamydia testing uptake between MSM and non-MSM participants across the three intervention arms.
Time Frame: During enrollment visit
Measure: Count of Participants; unit: Participants
Groups:
- Community-engaged Pay-It-Forward: Participants received free gonorrhea and chlamydia testing donated by previous participants and were offered an opportunity to make monetary and/or handwritten message donations to support other participants among MSM versus non-MSM.
- Standard Pay-It-Forward: Participants received free gonorrhea and chlamydia testing donated by previous participants and were offered an opportunity to make monetary donations to support other participants MSM versus non-MSM.
- Control: Participants received gonorrhea and chlamydia testing at an out-of-pocket cost of approximately $21 U.S.Dollars (USD) MSM versus non-MSM.
Arm/Group | Community-engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 400
Participants
  MSM | 194 | 193 | 1
  Non-MSM | 196 | 168 | 11
  Not Tested | 10 | 39 | 388
Statistical Analysis 1: Comparison: Community-engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; We anticipated a test uptake of 65% in the community-engaged pay-it-forward arm, 45% in the standard pay-it-forward arm, and 20% in the control among MSM and non-MSM participants; Test type: Other; p = 0.015, Generalized Estimating Equations; Difference in Probability Difference = -0.040, 95% CI [-0.073 to -0.008]

12. Other Pre Specified Outcome: Gonorrhea and Chlamydia Testing Uptake by Age Group
Description: Stratifies gonorrhea/chlamydia testing uptake between participants aged 30 years and below and those above 30 years across the three intervention arms.
Time Frame: During enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Community-engaged Pay-It-Forward | Standard Pay-It-Forward | Control
Number analyzed (Participants) | 400 | 400 | 400
Participants
  30 years and below | 143 | 178 | 4
  Above 30 years | 247 | 183 | 8
  Not Tested | 10 | 39 | 388
Statistical Analysis 1: Comparison: Community-engaged Pay-It-Forward vs Standard Pay-It-Forward vs Control; We anticipated a test uptake of 65% in the community-engaged pay-it-forward arm, 45% in the standard pay-it-forward arm, and 20% in the control among participants 30 years and below and those above 30 years; Test type: Other; p = 0.384, Generalized Estimating Equations; Difference in Probability Difference = 0.015, 95% CI [-0.019 to 0.049]

ADVERSE EVENTS:
Time Frame: Baseline through follow-up (an approximate total of 3 months)
Groups:
- Community Engaged Pay-it-forward: Participants received free gonorrhea and chlamydia testing donated by previous participants and were offered an opportunity to make monetary and/or handwritten message donations to support other participants.
- Control Arm: Participants received gonorrhea and chlamydia testing at an out-of-pocket cost of approximately $21 U.S. Dollars (USD).
Arm/Group | Community Engaged Pay-it-forward | Standard Pay-it-forward | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/400 | 0/400
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/400
Other Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/400

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT05723263/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Amended Study Protocol and Statistical Analysis Plan (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT05723263/Prot_SAP_003.pdf
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT05723263/ICF_000.pdf